CLINICAL TRIAL: NCT06464874
Title: Hybrid Versus Conventional Endoscopic Submucosal Dissection for Laterally Spreading Tumors (LSTs): A Retrospective Multicenter Study
Brief Title: Endoscopic Therapy for Laterally Spreading Tumors (LSTs)
Acronym: LST
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0444
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2020-05

CONDITIONS: To Compare the Efficacy and Safety of Hybrid ESD and ESD in the Treatment of Colorectal LST
Keywords: Colorectal adenoma；Laterally spreading tumors, Endoscopic submucosal dissection, Hybrid endoscopic submucosal dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional ESD: Submucosal injection of methylene blue solution at various sites was performed, followed by periphery incision using a dual knife. The submucosal injection was administered multiple times, followed by the utilization of an IT knife for submucosal separation and gradual excision of the lesion. In cases of significant bleeding at the wound site, electrocoagulation hemostatic forceps were employed for hemostasis.
  Interventions: Procedure: Conventional ESD
- hybrid ESD: The submucosal injection and circumferential incision of the Hybrid ESD were performed as described above. Subsequently, snaring was conducted post submucosal dissection utilizing a polypectomy snare for complete lesion removal. Careful attention was paid during excision to avoid muscle layer penetration and to control cutting speed in order to mitigate the potential for hemorrhage and perforation. The subsequent steps of the procedure closely followed the conventional ESD methodology outlined previously.
  Interventions: Procedure: Hybrid ESD

INTERVENTIONS:
Procedure: Conventional ESD — Conventional ESD is the most suitable method for total resection, especially for large lesions. This method can complete the resection of early gastrointestinal cancer and precancerous lesions, while maintaining the integrity of digestive tract anatomy and physiological function.The operation difficulty of this technique is high, the equipment requirements are high, the operation time is long, and the complication rate is closely related to the technical level of the operator.
  Groups: conventional ESD
Procedure: Hybrid ESD — Hybrid ESD is a better choice, but only can remove the lesion in one piece, but also has a lower technical difficulty than conventional ESD
  Groups: hybrid ESD

SUMMARY:
This study will retrospectively include LST patients who were admitted to 6 medical centers (The Second Affiliated Hospital, College of Medicine, Zhejiang University; The Affiliated Jinhua Hospital, Zhejiang University School of Medicine; First Affiliated Hospital of Huzhou University; The Second Hospital of Jiaxing; Jinhua People's Hospital; Lanxi People's Hospital) from 2020.05.01 to 2023.04.30 with the purpose of comparing the efficacy and safety of hybrid ESD and ESD in the treatment of colorectal LST. The complete resection rate, operation time, operation cost, intraoperative and postoperative complications of hybrid ESD and ESD LST will be compared. To provide strong evidence for the selection of endoscopic treatment strategies for LST.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* LST lesion diameter >1cm;
* Medical record data integrity

Exclusion Criteria:

* Pedicle lesions;
* Resection of residual lesions after endoscopic treatment;
* Advanced endoscopic imaging showed submucosal infiltrating lesions.
* The lesions are in patients with inflammatory bowel disease;
* Familial polyposis;
* Electrolyte abnormalities;
* Coagulation dysfunction;
* Pregnant or lactating patients;
* Taking nonsteroidal anti-inflammatory drugs or anticoagulants;
* A history of alcoholism;
* Severe organ failure;
* Medical records are incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involved a multicenter retrospective analysis of 890 consecutive patients with a colorectal LST > 10 millimeters who underwent endoscopic treatment at 6 medical centers (The Second Affiliated Hospital, College of Medicine, Zhejiang University; The Affiliated Jinhua Hospital, Zhejiang University School of Medicine; First Affiliated Hospital of Huzhou University; The Second Hospital of Jiaxing; Jinhua People's Hospital; Lanxi People's Hospital) between May 2020 and April 2023.
Sampling Method: Non-Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
complete resection rate | 2 weeks
  One-time complete excision

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided